CLINICAL TRIAL: NCT03004599
Title: Safety and Efficacy of SYM-SV/DS-002 in Patients With Severe Aortic Stenosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the business issues. Manufacturer has been acquired by other company.
Sponsor: Medico's Hirata Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH-P-002
Record Dates: First submitted 2016-12-09; First posted 2016-12-29 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Severe Aortic Stenosis
Keywords: Valvular Heart Disease; Critical Aortic Stenosis; Severe Aortic Stenosis; High Risk; Aortic Valve Replacement; Cardiovascular Disease; Aortic Stenosis; Heart Valve Therapy; Transcatheter; Transfemoral; TAVI; TAVR; ACURATE neo™ Aortic Bioprosthesis; ACURATE TF™ Transfemoral Delivery System
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Cardiovascular Diseases

ARMS (1):
- Transcatheter Aortic Valve Implantation (TAVI) (Other)
  Interventions: Device: SYM-SV-002 Aortic Bioprosthesis and SYM-DS-002 Transfemoral Delivery System

INTERVENTIONS:
Device: SYM-SV-002 Aortic Bioprosthesis and SYM-DS-002 Transfemoral Delivery System — Transcatheter Aortic Valve Implantation via Transfemoral Approach
  Other Names: ACURATE neo™ Aortic Bioprosthesis; ACURATE TF™ Transfemoral Delivery System

SUMMARY:
Safety and Efficacy of SYM-SV/DS-002 in Patients with Severe Aortic Stenosis

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of Transfemoral Transcatheter Aortic Valve Implantation using SYM-SV-002 Aortic Bioprosthesis and SYM-DS-002 Transfemoral Delivery System in patients presenting with symptomatic severe aortic stenosis and with difficulty to safely undergo conventional surgical aortic valve replacement (AVR)

ELIGIBILITY:
Inclusion Criteria:

1. At least one cardiologist and one cardiac surgeon agree that it is difficult for the patient to receive a surgical procedure due to medical factors such that the subject has various comorbidities and he/she is more likely to die or suffer from severe diseases than to have significant improvements by a surgical procedure.
2. Subject has senile degenerative aortic valve stenosis with:

   * mean gradient > 40 mmHg, or maximum jet velocity greater than 4.0 m/sec by either resting or dobutamine stress echocardiogram, or simultaneous pressure recordings at cardiac catheterization
   * AND an initial aortic valve area of ≤ 0.8 cm2 (or aortic valve area index ≤ 0.5 cm2/m2) by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization
3. Subject is symptomatic from his/her aortic valve stenosis (AS), as demonstrated by New York Heart Association (NYHA) Functional Class II or greater.
4. The subject has been informed of the nature of this trial, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site.
5. The subject or the subject's legal representative agrees to visit the site where he/she receives index procedure for all required post-procedure follow-ups.

Exclusion Criteria:

1. Evidence of an acute myocardial infarction ≤ 30 days (The procedure day is counted as day 0.) before the implant procedure
2. Any percutaneous coronary or peripheral interventional procedures, including placements of bare metal stents are performed within 30 days prior to the implant procedure, or any drug eluting stents are placed within 6 months (One month is counted as 30 days.) prior to the implant procedure
3. Untreated clinically significant coronary artery disease (CAD) requiring revascularization
4. Blood dyscrasias as defined:

   leukopenia (WBC < 1,000/mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy
5. Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support
6. Need for emergency surgery for any reason
7. Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% as measured by resting echocardiogram
8. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to the implant procedure (except mild TIA related to aortic stenosis)
9. End stage renal disease requiring chronic dialysis or serum creatinine > 3.0 mg/dL
10. Active Gastrointestinal (GI) bleeding within 3 months prior to the implant procedure
11. A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:

    * Aspirin
    * Heparin (HIT/HITTS)
    * Nitinol (titanium or nickel)
    * P2Y12 inhibitors (such as Ticlopidine etc.)
    * Contrast media
12. Ongoing sepsis, including active endocarditis
13. Subject refuses a blood transfusion
14. Life expectancy < 12 months due to associated non-cardiac comorbid conditions
15. Other medical, social, or psychological conditions that in the opinion of a principal investigator or sub-investigator precludes the subject from appropriate consent
16. Severe dementia (unable to provide informed consent for the treatment/procedure, unable to live an independent life outside of a chronic care facility, or expected to be fundamentally unable to undergo rehabilitation after the procedure, or unable to come to the site for follow-up visits)
17. Currently participating in other trials of investigational drugs or other investigational devices
18. Native aortic annulus size < 21 mm or > 27 mm per the baseline diagnostic imaging
19. Pre-existing prosthetic heart valve and / or prosthetic ring in any position
20. Mixed aortic valve disease (aortic stenosis and predominant aortic regurgitation (3-4+))
21. Moderate to severe (3-4+) or severe (4+) mitral regurgitation or severe (4+) tricuspid regurgitation
22. Moderate to severe mitral stenosis
23. Hypertrophic obstructive cardiomyopathy
24. New or untreated echocardiographic evidence of intracardiac mass, thrombus or vegetation
25. Congenital bicuspid or unicuspid valve verified by echocardiograph
26. Extreme eccentric calcification of the native aortic valve
27. Transesophageal echocardiogram (TEE) is contraindicated.
28. Scheduled surgical or percutaneous procedure to be performed prior to 1-month visit post-implant procedure
29. Hepatic failure (Child C or more)
30. Aortic or peripheral condition NOT appropriate for transfemoral implant due to the size, disease and degree of calcification or tortuosity of the aorta or ilio-femoral arteries
31. Thoracic or abdominal aortic aneurysm
32. Woman who is pregnant, breastfeeding or willing to become pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Survival rate | at 12 months post-procedure

SECONDARY OUTCOMES:
Occurrence rates of MACCE | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  MACCE is defined as a composite of:
  * All Cause Mortality
  * Myocardial infarction (MI)
  * All Stroke
  * Reintervention
Occurrence rates of individual MACCE components | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Individual MACCE components include:
  * All Cause Mortality
  * Myocardial infarction (MI)
  * All Stroke
  * Reintervention
Occurrence rates of Major Adverse Events (MAEs) | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  MAEs include:
  * MACCE
  * Acute Kidney Injury (AKI)
  * Cardiac Tamponade
  * Prosthetic Valve Dysfunction (PVD)
  * Cardiogenic Shock
  * Prosthetic Valve Endocarditis
  * Life-Threatening, Disabling or Major Bleeding
  * Major Vascular Complications
  * Cardiac Perforation
  * Device Migration/Valve Embolism
Occurrence rate of conduction disturbance requiring Permanent Pacemaker Implantation(PPI) | at 1 month, 6 month, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
Change in NYHA class from baseline | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
Change in distance walked during 6-Minute Walk Test (6MWT) from baseline | at 1 month and 12 month post-procedure
Change in QOL from baseline | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Kansas City Cardiomyopathy Questionnaire (KCCQ)
Change in QOL from baseline | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  SF-36
Echocardiographic assessment of valve performance | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Effective Orifice Area Index (EOAI)
Echocardiographic assessment of valve performance | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Mean gradient
Echocardiographic assessment of valve performance | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Degree of Aortic valve Regurgitation (AR) (Transvalvular and Paravalvular)
Echocardiographic assessment of valve performance | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Left ventricular ejection fraction (LVEF)
Device success | Number of days from admission to discharge (estimated to be at 7 days post-procedure on average)
  Device success is defined as that all of the following are achieved:
  * Successful vascular access
  * Successful delivery and deployment of the device
  * Successful retrieval of the delivery system
  * Correct position of the device in the proper anatomical location (placement in the aortic annulus with no impedance on device function)
  * Intended performance of the prosthetic heart valve is confirmed by echocardiography (defined as below):
  * No Patient-Prosthesis Mismatch (PPM) (EOAI >0.85cm2/m2)
  * And mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/sec,
  * And no moderate or severe prosthetic valve regurgitation
  * Only one valve implanted in the proper anatomical location
Procedural success | Number of days from admission to discharge (estimated to be at 7 days post-procedure on average)
  Procedural success is defined as that all of the following are achieved:
  * Achievement of the device success
  * Absence of in-hospital MACCE
Occurrence rate of Prosthetic Valve Dysfunction (PVD) | at 1 month, 6 months, 12 months, 2 years, 3 years, 4 years and 5 years post-procedure
  Prosthetic Valve Dysfunction (PVD) is defined as:
  * Aortic regurgitation (AR) reported as moderate or severe by echocardiography assessments
  * Significant aortic stenosis (AS) which meets one or more of the following by echocardiography assessments:
  * Peak velocity > 4 m/s
  * Mean gradient > 35 mmHg
  * Effective Orifice Area (EOA) < 0.8 cm2
  * TVIV1／TVIV2 < 0.25
Occurrence rate of clinical endpoints per VARC 2 | at 1 month post-procedure
  * Mortality
  * Stroke
  * Myocardial infarction (MI)
  * Bleeding complications
  * Acute kidney injury (AKI)
  * Vascular complications
  * Conduction disturbances and arrhythmia
  * Other TAVI-related complications

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Osaka University Hospital, Suita, Osaka
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo